CLINICAL TRIAL: NCT04099121
Title: Evaluation of 3D Ultrasound Vaginal Manometry for Estimating the Optimal Pessary Size for Patients With Pelvic Organ Prolapse
Brief Title: Evaluation of 3D Translabial Ultrasound Imaging for Pessary Size Estimation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: Cosm Medical Corp. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 6086
Record Dates: First submitted 2019-05-01; First posted 2019-09-23 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Prolapse
MeSH Terms: conditions — Prolapse | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Pelvic Organ Prolapse (Other): Patients who meet the inclusion criteria will be recruited. Ultrasound images of the pelvic floor and vaginal cavity will be analyzed to predict pessary size and type. This will be compared against the pessary size and type being used already by the patient.
  Interventions: Device: Ultrasound Imaging

INTERVENTIONS:
Device: Ultrasound Imaging — 3D ultrasound of the pelvic floor and vaginal cavity will be obtained by using a commercial ultrasound system.

SUMMARY:
Symptoms of female pelvic floor dysfunction, such as incontinence and pelvic organ prolapse, can be alleviated by using pessaries, which are passive medical devices that are inserted in the vagina to support the pelvic organs. Currently, pessaries are fit through trial and error after manual examination, the accuracy of which depends on the physician's expertise level.

The objective of this study is to evaluate the feasibility of using 3D translabial ultrasound imaging of the vagina at various distension volumes to predict the pessary size for successful fit. Ultrasound images will be obtained using commercially available 3D ultrasound probes (Philips, Netherlands), as well as a commercially available 2D ultrasound probe (Philips, Netherlands), which is linearly scanned to capture a 3D volume. The linear scanning will be performed by attaching the 2D probe to a motorized hand-held scanner, which is used to tilt and move the probe to acquire images. Please note that the hand-held scanner does not come in contact with the patient. To distend the vagina, a sterile bag is inserted in the vagina and gradually filled with water using a commercially available urodynamic system (Laborie, Canada) until the vaginal capacity is reached, without causing any discomfort to the patient. This image acquisition technique, previously reported in the literature, is referred to as 3D ultrasound vaginal manometry in this study.

To achieve the objective of this project, 35 pelvic organ prolapse patients, who (i) are current pessary users, (ii) can perform self-care of the pessary, and (iii) can provide informed consent, will be invited to participate in the study. Patients will be asked to remove their pessary prior to ultrasound imaging. Then, 3D ultrasound vaginal manometry will be performed, using the technique described above. Ultrasound images will be analyzed once data acquisition is completed. The size of the pessary estimated from ultrasound images will be compared with the actual pessary size used by the patient.

ELIGIBILITY:
Inclusion Criteria:

* Current pessary users (> 6 months) who have no pessary related complication, including discomfort, repeated vaginal bleeding, and pessary extrusion
* Are able to provide informed consent
* Can perform self-care, i.e. removing and inserting the pessary themselves
* Are willing to remove their pessary 2 days before the ultrasound examination date.

Exclusion Criteria:

* Inability to give informed consent
* Inability to communicate with the person performing the consent and the sonographer performing ultrasound scanning
* History of pelvic radiation or surgery, (including hysterectomy)
* Using pessaries other than ring, incontinence dish, donut, Shaatz, Marland, or Gellhorn.
* Inability to perform the Valsalva maneuver or pelvic floor contraction
* Restricted mobility that prevents them from ambulating to assess the comfort level of the pessary during the initial pessary fitting visit.
* Lack of sensation at the pelvic floor.
* Being pregnant at the time of the examination.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pelvic organ prolapse only occurs in females.
Enrollment: 24 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
FEASIBILITY: The predicted pessary size | Up to 3 months following data collection
  The predicted pessary size in cubic mm will be compared with the actual size of the pessary used by the patient
FEASIBILITY: The predicted pessary shape | Up to 3 months following data collection
  The predicted pessary shape will be compared with the actual shape of the pessary used by the patient by calculating the DICE coefficient.

CONTACTS AND LOCATIONS:
Locations (1):
- Victoria Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Data will be de-identified, and only the aggregate results will be used for publication. Patient information will not be made public or shared with researchers outside of the study team.